CLINICAL TRIAL: NCT06064838
Title: Effects of Cacao Flavonoids in Long COVID-19 Patients with Chronic Fatigue (FLALOC)
Brief Title: Effects of Cacao Flavonoids in Long COVID-19 Patients (FLALOC)
Acronym: FLALOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guillermo Ceballos Reyes (Other)
Collaborators: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Sponsor-Investigator, Guillermo Ceballos Reyes, Professor, National Polytechnic Institute, Mexico
Organization: National Polytechnic Institute, Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FLALOC
Record Dates: First submitted 2023-10-02; First posted 2023-10-03 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Long Covid19; Fatigue Syndrome, Chronic
Keywords: flavonoids; post-covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic | interventions — Flavonoids; Chocolate

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled clinical trial will be conducted at the specialty clinic Indianilla in Mexico City, during the period from August 2023 to September 2024 with post-covid patients with chronic fatigue.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flavonoids (Experimental): Capsules with 500mg of cacao flavonoids, twice a day for 90 days
  Interventions: Dietary Supplement: Flavonoids
- Placebo (Placebo Comparator): Capsules with 500mg of excipients, twice a day for 90 days
  Interventions: Dietary Supplement: Flavonoids

INTERVENTIONS:
Dietary Supplement: Flavonoids — 1 capsule every 12h for 90 days
  Other Names: Cacao and Health EC-Fitness

SUMMARY:
The study use a triple blind, placebo-controlled design enrolling male and female subjects between 30-70 yo to evaluate the effect of daily consumption of a cacao supplement on inflammation, endothelial damage, handgrip strength, fatigue scale and quality of life.

DETAILED DESCRIPTION:
The study use a triple blind, placebo-controlled design enrolling male and female subjects between 30-70 yo distributed homogeneously at random in two groups: the control group (Placebo) and the intervention group (Cacao Flavonoids) both groups affected for 90 days.

The variables to consider will be: Interleukins (IL-1b, IL-6), Tumoral Necrosis Factor alpha (TNF-α) and syndecan-1.

For physical performance is evaluated the handgrip strength. The investigators also assessed quality of life using the Health Related QoL (EQ-5D) questionnaire, and the numerical fatigue rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID-19 patients, at least 6 months after symptom onset
* Chronic fatigue

Exclusion Criteria:

* Allergy or intolerance caused by active ingredients
* Pregnancy or lactation
* BMI >35
* chronic liver disease
* chronic kidney disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Interleukin-1b | At 0 and 90 day
  Plasmatic concentration
Interleukin-6 | At 0 and 90 day
  Plasmatic concentration
TNF-alpha | At 0 and 90 day
  Plasmatic concentration
Syndecan-1 | At 0 and 90 day
  Plasmatic concentration

SECONDARY OUTCOMES:
EQ-5D questionnaire | At 0 and 90 day
  Self-administered health index that explores five domains
Analog Visual Scale | At 0 and 90 day
  Use of a Analog Visual Scale to measure the quality of life, graded 0 (worst) to 100 (best) for the perception of wellbeing.
Numerical fatigue rating scale | At 0 and 90 day
  fatigue rating scale graded 0 (best) to 100 (worst)
Handgrip strength | At 0 and 90 day
  Measures static force in kilograms that the hand can squeeze around a dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- C.E. Indianilla, Mexico City, Mexico City, Mexico